CLINICAL TRIAL: NCT02067936
Title: Walking the Isobole of Drug Interaction: Comparison of Hemodynamic Effects, Cerebral and Tissue Oxygenation for 4 Equipotent Combinations of Propofol and Remifentanil
Brief Title: Walking the Isobole of Drug Interaction
Acronym: Walibi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Hugo E.M.Vereecke, Dr., University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: WALIBI-001
Record Dates: First submitted 2014-02-03; First posted 2014-02-20 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Hemodynamic Instability; Disorder of Oxygen Transport; Interaction; Anesthesia
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A propofol + remifentanil (Active Comparator): Propofol highest dose, remifentanil lowest dose, TOL 90% according to Bouillon model
  Interventions: Drug: Group A propofol + remifentanil
- Group B propofol + remifentanil (Active Comparator): Propofol intermediate high, remifentanil intermediate low, TOL90% according to the Bouillon Model
  Interventions: Drug: Group B propofol + remifentanil
- Group C propofol + remifentanil (Active Comparator): propofol intermediate low+ remifentanil intermediate high: TOL 90% according to the Bouillon interaction model
  Interventions: Drug: Group C propofol + remifentanil
- group D propofol + remifentanil (Active Comparator): propofol lowest dose+ remifentanil highest dose: TOL 90% according to the Bouillon model
  Interventions: Drug: group D propofol + remifentanil

INTERVENTIONS:
Drug: Group A propofol + remifentanil — Predicted TOL90% according to Bouillon model
  Other Names: propofol highest dose + remifentanil lowest dose
  Arms: Group A propofol + remifentanil
Drug: Group B propofol + remifentanil — TOL 90% according to the Bouillon interaction model
  Other Names: Propofol intermediate high+ remifentanil intermediate low
  Arms: Group B propofol + remifentanil
Drug: Group C propofol + remifentanil — TOL 90% according to the Bouillon interaction model
  Other Names: propofol intermediate low+remifentanil intermediate high
  Arms: Group C propofol + remifentanil
Drug: group D propofol + remifentanil — TOL 90% according to the Bouillon interaction model
  Other Names: Propofol lowest dose+ remifentanil highest
  Arms: group D propofol + remifentanil

SUMMARY:
The investigators study whether four equipotent combinations of propofol and remifentanil (as predicted by interaction models for "tolerance of laryngoscopy") result in identical haemodynamic conditions, independent of their relative different balance between the concentration of propofol and remifentanil.

DETAILED DESCRIPTION:
In anesthesia, the synergistic interaction between hypnotics and opioids is applied daily to give adequate anesthesia and analgesia at significantly lower doses compared with the ones needed if only one drug was given to reach the same effect. A lot of research has been done to quantify these interactions with a focus on the desired effects (Tolerance of laryngoscopy, tolerance of shake and shout etc...), but the simultaneous interaction on the unwanted side effects is less well described. The response surface model of Bouillon et al. and other models predict combinations of propofol and remifentanil effect-site concentrations that lead to an equipotent desired effect. Due to the availability of the models, the anesthesiologists now could use the knowledge on interactions to target specific effects more accurately, using predefined equipotent combinations of drugs: for instance, a desirable 90% probability of tolerance of laryngoscopy (TOL90) in the population can be reached through either a high propofol/low remifentanil combination, but equally well through a low propofol-high remifentanil combination.

However, at this time it is not known whether some of the combinations of propofol and remifentanil have a favorable hemodynamic stability compared to other equipotent combinations. The researcher in this study want to determine whether equipotent combinations of remifentanil and propofol (all deliberately selected to evoke 90% probability of "tolerance to laryngoscopy"), result in different effects on the undesired side effects of anesthetics, such as hemodynamic instability (hypotension, changes in heart rate or cardiac output), decreases in cerebral or tissue oxygenation (both measured with near infrared spectroscopy).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* General anesthesia required for the procedure
* Age: 18 years and older
* American Society of Anesthesiologists (ASA) physical status I to III

Exclusion Criteria:

* Refusal to participate in this study
* Contra-indications for the use of propofol or remifentanil
* BMI > 35 kg/m2
* Central nervous system disorders (i.e. cerebrovascular accident, dementia, seizures, psychiatric disorders)
* Relevant hepatic disease (Child B or higher)
* Regular use of medication that affects the central nervous system (i.e. benzodiazepines, antidepressants, antipsychotics, antiepileptic drugs)
* Use of alpha-agonists or beta-blockers
* Overt signs of alcohol abuse
* Use of preoperative benzodiazepines (on the day of the study)
* Beta blockers eye drips
* Overt signs of Drugs abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure | From start drug till intubation which will take on average 15 minutes of measurement
  Continuously stored on a laptop (systolic, diastolic and mean blood pressure over time) using a Philips Non Invasive Blood Pressure measurements every minute and a Nexfin monitor (continuous non invasive blood pressure measurement)

SECONDARY OUTCOMES:
Electro Encephalographic derived indices of anesthetic depth | From start first drug till intubation, which will take on average 15 minutes of measurement
  Bispectral index, Wavelet Transformation (WAV) index, Quantium Consciousness Index (qCON), Quantium Nociception Index (qNOX) to observe whether multiple electroencephalographic derived depth of anesthesia indices indicate the same equipotent effect in all 4 groups. All these measures are unitless values that range between 100 (for a fully responsive condition) and 0 (for a fully unresponsive condition). All these measures are extracted from the same frontal electroencephalogram but use different composite mathematical algorithms to translate the cortical state in numbers. We want to observe whether these composite algorithms measure consistent behavior between groups. This outcome is mainly ment as hypothesis generating for future research.
Cerebral and tissue oxygenation | From start drug till intubation, which will take on average 15 minutes of measurement
  Continuously stored oxygenation saturation measured in tissue and cerebral cortex as measured by Near Infrared Spectrum Analysis (Forsyth monitor) and Inspectra monitor. Comparing differences between 4 groups with ANOVA.
Heart rate | From start first drug till intubation, which will take on average 15 minutes of measurement
  Difference in median/mean heart rate to determine differences between 4 groups with ANOVA.
Probability of tolerance to laryngoscopy | one minute before laryngoscopy till three minutes after
  During pharmacological steady state of propofol/remifentanil, a laryngoscopy will be performed by one researcher and response or tolerance of the stimulus will be observed. A positive response will be defined as any somatic movement, swallowing or coughing during three minutes after laryngoscopy was applied. Also a increase in heart rate or systolic blood pressure of more than 20% from baseline values (one minute before laryngoscopy) will be defined as a positive response. Through PROBIT analysis we can plot the probability of response to laryngoscopy (%) as a function of respectively propofol or remifentanil drug concentrations.
Cardiac index | From start first drug till intubation, which will take on average 15 minutes of measurement
  Non invasive estimation of Cardiac output and Cardiac index patterns through the Nexfin monitor. Determine the differences between groups through ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo EM Vereecke, MD, PhD, Principal Investigator — University Hospital Medical center, university of groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands